CLINICAL TRIAL: NCT06971588
Title: The Role of Music in Enhancing Attention During Visual Field Exams for Pediatric Glaucoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB00484910
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
Keywords: Pediatric; Glaucoma; Music; Research; Ophthalmology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: The study will involve the child being randomized to a control and experimental group, and about 2 weeks after the initial test, they will be asked to come in and take part in the alternate study group. During the control visit, the child will take the visual field exam as they would in their routine care.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (first) (Experimental): This arm will involve the use of music during their initial VFE, and then they will take part in the non-music group during their second visit.
  Interventions: Other: Music intervention
- Non-Music Group (first) (Experimental): This arm will involve the completion of the VFE with no music first, and then they will crossover and complete the arm involving the use of music during the visual field exam.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — The intervention will involve patient-chosen music.

SUMMARY:
The goal of the study is to see if the use of music improves attention during visual field exams for pediatric glaucoma patients.

DETAILED DESCRIPTION:
This study aims to determine if music can be used as an intervention to improve attention and quality of results in pediatric glaucoma patients taking visual field exams. The investigators also want to determine the most effective method and type of music by which it can be implemented into the test to improve patient experience and results. If there is an improvement, it will benefit the patient and the provider in administering the test and the utility of the results.

To that end, patients between the ages of 8-17 with Glaucoma or glaucoma suspect diagnosis will be recruited from the clinic with consent from their parents and assent from the patient to participate in the study. They will come in on two scheduled dates after being randomized to either a control or experimental group. On the first date, the participants assigned to the control group will complete the Visual Field Exams (VFE) without music, and the experimental group will listen to music and complete a pre and posttest survey regarding test taking experience. On the second date, the groups will switch and the participant will complete the other part of the study. Results will then be analyzed and compared between the groups and previous results.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma or glaucoma suspect

Exclusion Criteria:

* Post operative patient
* Non English speaking

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of False Positives On VFE | Baseline, Follow-up visit up to 4 weeks
  This outcome measurement will be used to assess reliability by seeing how often the patients were responding to stimuli that weren't present during the VFE. Assessment will be done by the physician after completion of the VFE by patient which takes about 10 minutes.
Number of False Negatives On VFE | Baseline, Follow-up visit up to 4 weeks
  This measurement is a reliability tool to see if the patient missed any stimuli during VFE. Assessment will be done by the physician after completion of the VFE by patient which takes about 10 minutes.
Number of Fixation Losses on VFE | Baseline, Follow-up visit up to 4 weeks
  This will evaluate any gaze deviation by the patient during VFE as a marker of inattention and test reliability. Assessment will be done by the physician after completion of the VFE by patient which takes about 10 minutes.
Test Duration (minutes) On VFE | Baseline, Follow-up visit up to 4 weeks
  This will evaluate the length of the test as a marker for inattention and reliability if patient takes longer to complete the exam in one group or the other. Assessment will be done by the physician after completion of the VFE by patient which takes about 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Kraus, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muralidharan S, Ichhpujani P, Bhartiya S, Singh RB. Eye-tunes: role of music in ophthalmology and vision sciences. Ther Adv Ophthalmol. 2021 Sep 2;13:25158414211040890. doi: 10.1177/25158414211040890. eCollection 2021 Jan-Dec. PMID 34497975
- [Background] Blood AJ, Zatorre RJ. Intensely pleasurable responses to music correlate with activity in brain regions implicated in reward and emotion. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11818-23. doi: 10.1073/pnas.191355898. PMID 11573015
- See also: Baldwin, M., & Lewis, R. (2017). Positive valence music restores executive control over sustained attention. PLOS ONE, 12(11), e0186231. https://doi.org/10.1371/journal.pone.0186231 — https://doi.org/10.1371/journal.pone.0186231